CLINICAL TRIAL: NCT04472403
Title: Efficacy and Safety of Platinum Plus Continuous Intravenous Infused 5-Fluorouracil With Low Dose and Long Term Versus Other Platinum-Based Chemotherapy in Metastatic Nasopharyngeal Carcinoma: A Case-Cohort Study
Brief Title: Platinum Plus Low-dose Long-term Continuous Intravenous Infused 5-Fluorouracil in Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Other Study IDs: B2019-201-01
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Nasopharyngeal Carcinoma; Metastasis; Chemotherapy; Survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PFLL Group: Patients were treated with PFLL regimen: 5-fluorouracil intravenous infusion at 200mg/m2/d for 30 continuous days and intravenous infusion of platinum (cisplatin 70 mg/m2 or nedaplatin 80/m2 or lobaplatin 30 mg/m2) on day 1 and day 28, every 60 days.
  Local treatment, molecular-targeted or immune checkpoint therapy, and supportive treatment were allowed.
- Non-PFLL Group: Patients were treated with other platinum-based chemotherapy every 21 days including:
  PF regimen: 5-fluorouracil at a dose of 1,000 mg/m2 daily by continuous intravenous infusion on days 1-4 and intravenous infusion of cisplatin at a dose of 80 mg/m2 on day 1.
  GP regimen: gemcitabine at a dose of 1,000 mg/m2 by intravenous infusion on days 1, 8, and intravenous infusion of cisplatin at a dose of 80 mg/m2 on day 1.
  TP regimen: paclitaxel intravenous infusion at a dose of 175 mg/m2 or docetaxel at a dose of 75 mg/m2 on day 1 and intravenous infusion of cisplatin at a dose of 75 mg/m2 on day 1.
  TPF regimen: paclitaxel intravenous infusion at a dose of 175 mg/m2 or docetaxel at a dose of 75 mg/m2 on day 1; cisplatin intravenous infusion at a dose of 75 mg/m2 on day 1 and continuous intravenous infusion of 5-FU at a dose of 750 mg/m2 daily on days 1-5.
  Local treatment, molecular-targeted or immune checkpoint therapy, and supportive treatment were allowed.

SUMMARY:
The treatment of distant metastasis is a key challenge for nasopharyngeal carcinoma because of poor outcomes, among which, chemotherapy is the cornerstone. However, many studies reported the use of different chemotherapy regimens to prolong the survival of metastatic nasopharyngeal carcinoma, while few of them focused on how to reduce the side effects of chemotherapy or improve the life quality of patients. Thus, we sought to find an efficient chemotherapy regimen with high tolerance according to the characteristics of chemotherapy drugs, that is, to explore the efficacy and safety of platinum plus 5-fluorouracil with continuous intravenous infusion at a low dose for a long term.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a malignant tumor of the nasopharyngeal epithelium with high sensitivity to ionizing radiation. With the use of intensive chemoradiotherapy, excellent treatment outcomes can be achieved for local control, but disease failure was observed in approximately 20% of patients. Moreover, approximately 10% of newly diagnosed patients diagnosed with metastasis, resulting in about 30% of NPC patients will present with either synchronous or metachronous metastasis in total.

Chemotherapy is the cornerstone of the treatment of metastatic NPC. Many studies were aimed at the systemic treatment of metastatic NPC, but most of them were retrospective studies or phase II trials with small samples. The outcome of metastatic NPC is poor with a median OS of about 20 months. Platinum-containing doublet chemotherapy is generally regarded as the standard treatment for metastatic NPC. After a multicenter phase III randomized clinical trial was published in 2016, gemcitabine plus cisplatin is recommended, however, less than 60% of patients could complete the treatment in the trail. Finding a proper regimen with promising efficacy results as well as high tolerance is still a big challenge.

Cisplatin plus 5-fluorouracil (PF) is a classical regimen widely used in metastatic NPC. The continuous infusion of 5-fluorouracil with low dose was investigated in esophagus carcinoma, rectal carcinoma and prostate carcinoma with encouraging outcome and acceptable toxicity. Whereas, data of platinum-containing chemotherapy with low-dose continuous infused 5-fluorouracil in metastatic NPC was absent. In this study, we aimed to investigate the antitumor activity of platinum plus low-dose long-term continuous intravenous infused 5-fluorouracil (PFLL).

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal carcinoma diagnosed by pathology or cytology
* Distant metastasis confirmed by Radiographic assessments or pathology.
* Patients ever received systemic chemotherapy.

Exclusion Criteria:

* Age <18 or >70 years old
* Pathologic type unknown or except type I-III of World Health Organization classification
* Never underwent platinum-based chemotherapy
* Lack of information about T classification and N classification when metastasis
* Lost follow-up within one month from the start of treatment for metastasis
* Without other malignances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients involved in our study were patients who had histologically or cytologically confirmed NPC with diagnosed distant metastasis during 2006-2017 and receiving treatment in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years after diagnosis of metastasis
  The period until death is detected.
5-year subsequent-line treatment-free survival | 5 years after the start of the first-line treatment
  The period until earliest of the start date of subsequent-line treatment or death is detected.
5-year survival without symptoms and toxicity | 5 years after diagnosis of metastasis
  The period until any events (death or disease progression or ≥grade 3 chemotherapy-related haematological toxicity) is detected.

SECONDARY OUTCOMES:
Haematological toxicity | From the start of the first-line treatment, evaluation was performed every cycle during the treatment and then every 3-6 months after the completion of the treatment, up to the start of subsequent-line treatment or death or 5 years.
  The incidence of myelosuppression

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China